CLINICAL TRIAL: NCT04653051
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the DVR Plating System (Implant and Instrumentation) - A Retrospective Consecutive Series Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits of the DVR Plating System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-14T
Record Dates: First submitted 2020-11-19; First posted 2020-12-04 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Distal Radius Fracture; Distal Ulna Fracture; Osteotomy
Keywords: Medical Device; Performance; Safety; Clinical Benefits; Post-Market Clinical Follow-Up Study
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received DVR Plating System

SUMMARY:
The study is a single-center, retrospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to confirm safety, performance and clinical benefits of the DVR Plates. The primary objective is the assessment of performance by analyzing fracture healing. The secondary objective is the assessment of safety by recording and analyzing the incidence and frequency of complications and adverse events. Patients' outcomes will also be assessed.

DETAILED DESCRIPTION:
The DVR plating system in this study includes the DVR Crosslock Distal Radial Plate, the DVR Volar Rim Plate and the DVR Wrist Plates.

One site will be involved in this study. The aim is to include a total of 112 consecutive series patients treated between 2014 and 2018. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop, intraop, immediate post-op and last consultation visit will be available in medical notes and collected retrospectively. During a follow up phone call the patient will be asked to complete a patient questionnaire and a question on his/her wrist function. In addition, any complications since the last consultation visit at the clinic, information about and treatment of the complications will also be collected over the phone.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have been implanted with one of the DVR Plates according to the approved indications.

Exclusion Criteria:

* Off-label use.
* Cases where there is an active infection.
* Conditions which tend to retard healing such as, blood supply limitations, previous infections, etc.
* Insufficient quantity or quality of bone to permit stabilization of the fracture.
* Conditions that restrict the patient's ability or willingness to follow postoperative instructions during the healing process.
* Foreign body sensitivity - where material sensitivity is suspected, appropriate tests should be conducted and sensitivity ruled out prior to implantations.
* Cases where the implant(s) would cross open epiphyseal plates in skeletally immature patients.
* Cases with malignant primary or metastatic tumors which preclude adequate bone support or screw fixations, unless supplemental fixation or stabilization methods are utilized.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients must have received one of the DVR Plates and who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Southampton General Hospital, Southampton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Southampton General Hospital
Pre-assignment Details: 191 consecutive patients were identified at the Southampton General Hospital. 11 patients died or moved out of the area so they could not be enrolled. So 180 patients were contacted and were asked to consider their study participation. 69 patients were either not reachable within three attempts or declined study participation leaving us with 111 patients enrolled into this study.
Units Other Than Participants: cases
Groups:
- DVR Plating System: Single study patient cohort, including 111 participants (115 cases) who meet the inclusion/exclusion criteria and who received the DVR Plating System and have a mean follow-up of 3.8 years
Period: Last Consultation Visit at the Hospital
Arm/Group | DVR Plating System
Started | 111; 115 cases
Completed | 111; 115 cases
Not Completed | 0; 0 cases
Period: Follow-up Phone Call
Arm/Group | DVR Plating System
Started | 111; 114 cases
Completed | 111; 114 cases (One patient received two plates and one plate needed to be explanted before the follow.up phone call. Therefore this case, is not considered here)
Not Completed | 0; 0 cases

BASELINE CHARACTERISTICS:
Population: This is a retrospective study meaning that retrospective data from preoperative, operative, immediate postoperative and last consultation visit was collected from patients' charts that have been operated in the past. Due to this retrospective design of the study the retrieval of demographic information from past medical records was not always possible as some medical records did not contain all information.
Units Other Than Participants: cases
Groups:
- Subjects Received DVR Plating System: Single study patient cohort, including 111 participants (115 cases) who meet the inclusion/exclusion criteria and who received the DVR Plating System and have a mean follow-up of 3.8 years
Arm/Group | Subjects Received DVR Plating System
Number analyzed (Participants) | 111
Number analyzed (cases) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years
  years | 60.1 (18.5)
Sex: Female, Male [Count of Units; unit: cases]
  Female | 76
  Male | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Units; unit: cases]
  United Kingdom | 115
Weight, Continuous [Mean (Standard Deviation); unit: Kg] — Population: As the retrieval of the demographic data was not always possible the number of cases for the weight differs from the total amount of cases.
  Kg
    number analyzed (Participants) | 64
    number analyzed (cases) | 64
    (all) | 73.8 (17.8)
Height, Continuous [Mean (Standard Deviation); unit: cm] — Population: As the retrieval of the demographic data was not always possible the number of cases for the height differs from the total amount of cases.
  cm
    number analyzed (Participants) | 52
    number analyzed (cases) | 52
    (all) | 165.8 (16.2)
Body Mass Index, Continuous [Mean (Standard Deviation); unit: Kg/m^2] — Population: As the retrieval of the demographic data was not always possible the number of cases for the body mass index differs from the total amount of cases.
  Kg/m^2
    number analyzed (Participants) | 49
    number analyzed (cases) | 49
    (all) | 26.3 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Fracture Healing Based on Clinical Measures and X-rays
Description: Fracture healing will be evaluated by x-rays and clinical measures (no pain at fracture site)
Time Frame: Mean time of 3.8 years after the surgery
Measure: Count of Units; unit: cases
Units Other Than Participants: cases
Arm/Group | DVR Plating System
Number analyzed (Participants) | 111
Number analyzed (cases) | 115
cases
  X-ray Evaluation: Fracture/Osteotomy healed | 103
  X-ray Evaluation: Fracture/Osteotomy not healed | 2
  X-ray Evaluation: Fracture/Osteotomy healing not assessed | 10
  Clinical Evaluation: Fracture/Osteotomy healed | 114
  Clinical Evaluation: Fracture/Osteotomy not healed | 0
  Clinical Evaluation: Fracture/Osteotomy healing not assessed | 1

2. Secondary Outcome: Product Safety Based on Complications
Description: Safety will be assessed by recording and analyzing the incidence and frequency of complications. The complications are classified per ISO 14155 Definitions: Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), Serious Adverse Device Effects (SADEs).
  .
Time Frame: Mean time of 3.8 years after surgery
Population: complications [Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Device Effects (ADEs), Serious Adverse Device Effects (SADEs)] that occurred in the study cohort during the time of the study
Measure: Count of Units; unit: complications classified per ISO14155
Units Other Than Participants: complications classified per ISO14155
Arm/Group | DVR Plating System
Number analyzed (Participants) | 111
Number analyzed (complications classified per ISO14155) | 92
complications classified per ISO14155
  Adverse Events (AEs) | 77
  Serious Adverse Events (SAEs) | 4
  Adverse Device Effects (ADEs) | 11
  Serious Adverse Device Effects (SADEs) | 0

3. Secondary Outcome: Patient's Outcomes Were Also Assessed
Description: Patients were asked to complete a patient questionnaire (Patient-Rated Wrist Evaluation Score- PRWE)* and a question on their wrist function**
  * the PRWE is a self-administered, patient-specific questionnaire that consists of 15 items. It was designed to measure wrist pain and disability in activities of daily living, and consists of two subscales: pain and function. A score of 100 represents the worst functional score, whereas 0 represents no disability
  ** Patient reported outcome: assessment of fractured wrist comparing to before injury on a scale from 0 to 10, 0 being worst imaginable, and 10 being as good as before the injury.
Time Frame: Mean time of 3.8 years after surgery
Population: In a case the General Wrist Function could not be assessed as the patient is suffering from Kienbock's disease and is experiencing a lot of pain, therefore the General Wrist Function is calculated for 113 cases.
Measure: Mean (Standard Deviation); unit: cases
Units Other Than Participants: cases
Arm/Group | DVR Plating System
Number analyzed (Participants) | 111
Number analyzed (cases) | 114
cases
  PRWE Score | 12.8 (17.9)
  General Wrist Function: number analyzed (Participants) | 110
  General Wrist Function: number analyzed (cases) | 113
  General Wrist Function | 8.0 (2.1)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events from the date each subject was implanted up to 3.8 years after surgery, when the last follow-up was performed and patients completed the study.
Description: Adverse Event Reporting Description Adverse events were collected in an excel database on the tab of Adverse events, which gathers information on the date of occurrence, the nature of the adverse event, whether the device was involved, which treatment was used and the treatment outcome.
Groups:
- 111 Subjects Received DVR Plating System With a Mean Follow-up of 3.8 Years: Single study patient cohort, including 111 participants (115 patients) who meet the inclusion/exclusion criteria and who received the DVR Plating System
Arm/Group | 111 Subjects Received DVR Plating System With a Mean Follow-up of 3.8 Years
All-Cause Mortality (participants affected / at risk) | 0/111
Serious Adverse Events (participants affected / at risk) | 4/111
Other Adverse Events (participants affected / at risk) | 59/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 111 Subjects Received DVR Plating System With a Mean Follow-up of 3.8 Years (N=111)
Altered sensation of the median nerve (Nervous system disorders) | 1 (1) — Altered sensation of the median nerve
Car accident (Injury, poisoning and procedural complications) | 1 (1) — Fracture of ribs and hip due to a car accident
Reduced mobility (Musculoskeletal and connective tissue disorders) | 1 (1) — Reduced mobility, as patient unable to use the left thumb which heavily impacts the ability to perform any task with left hand - patient reported this was due to a ruptured tendon as a result of plaster cast
Kienbock's disease (Vascular disorders) | 1 (1) — Patient is experiencing ongoing significant pain due to Kienbock's disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 111 Subjects Received DVR Plating System With a Mean Follow-up of 3.8 Years (N=111)
Pain due to altered sensation (Nervous system disorders) | 1 (1) — Patient experiences shooting pains in hand. Surgery wasn't offered as wasn't thought to improve outcome. Subject is seeing independent specialist and was discharged from clinic.
Plate removal (Nervous system disorders) | 1 (1) — Patient had wrist plate removed due to "rubbing against nerve-screw was pressing against skin". Patient pointed out a small lump on the radial border of wrist which is quite tender and possibilities this may be a screw.
Shoulder/ arm pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient received epidural injection for trapped nerve/shoulder/arm pain
Pain in wrist (Musculoskeletal and connective tissue disorders) | 3 (3) — 1. Ongoing pain in wrist - described as "mild" 2. Regular ongoing pain in wrist since operation when performing tasks with affected wrist 3. Significant pain when using wrist and unable to straighten ring and little finger also weakness in wrist
Loose screw (Product Issues) | 1 (1) — Patient said a screw was "loose" according to the x-rays during clinic appointment - has not caused any issues
Stiffness and pain (Musculoskeletal and connective tissue disorders) | 3 (3) — 1. Stiffness and pain causing difficulty moving the hand-removal of used K-wires 2. Shoulder pain and stiffness 3. Stiffness in wrist
Shooting spasm pains (Musculoskeletal and connective tissue disorders) | 2 (2) — Experiences shooting spasm pains down arm and wrist - especially when using wrist a lot during working. Pain is not bad enough to stop subject from doing anything. 2- Patient experiences very occasional sudden shooting pain - no clear cause
Rotator cuff impingement (Nervous system disorders) | 1 (1) — Rotator cuff impingement with long head of biceps medialisation. Severe stiffness due to multiple injuries and prolonged reduced mobilization.
Collapsed joint line (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 2 (2) — 1. Patient reported there was a gap between the bones in wrist. Pain when using wrist and a 'clunking' 2. Pain is flaring up from time to time. Very active and pain mostly occurs recently during activities like climbing Nothing to note in X-Rays
Mild ache (Musculoskeletal and connective tissue disorders) | 2 (2) — 1. Patient experiences 'clicking' in wrist when moving with a "mild ache" 2. Patient experiences occasional mild pain when it's cold
Intermittent pain and instability (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient experiences intermittent pain in wrist and mentioned experiencing ongoing instability and it has some deformity -There was pre-existing instability of the DRUJ therefore the complication is unrelated to the device.
Lower Respiratory Tract Infection (LRTI) (Infections and infestations) | 1 (1) — Patient developed a LRTI post op and was given a course of antibiotics - extended hospital stay
Arthritis (Immune system disorders) | 4 (4) — 1. Reduced wrist function and occasional pain due to ongoing arthritis 2. Patient developed arthritis in wrist 3. Arthritis in wrist -pain, mostly in cold weather. Post-OP onset 4. Arthritis in fingers- regular ongoing pain in wrist
Low wrist function (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient attributed lower rated wrist function due to "stiff fingers"- unable to make a fist with left hand
Additional fall (Injury, poisoning and procedural complications) | 3 (3) — 1. Fall-no fracture but ligaments in arm/shoulder injured- pain affects wrist function 2. Fall, mobilizing with crutches-numbness in thumb and tip of little finger-reduced finger mobility 3. Patient had a subsequent fall, thumb injured- ongoing pain
Discomfort and pain (Product Issues) | 1 (1) — 1- Patient experienced discomfort and pain following operation. Shooting pain into ring and little finger, reduced grip and trouble rotating wrist
Polytrauma (Injury, poisoning and procedural complications) | 6 (6) — Polytrauma - long hospital stay
Aching and pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Subject experiences aching and some pain depending on the weather - affects subject intermittently
Plate removal (Product Issues) | 3 (3) — 1. Ongoing pain and eventually had metalwork removed 2. Pain caused plate removal 3. Ulna plate fixation failed in osteoporotic bone causing need for revision ulna fixation
Long recovery (Musculoskeletal and connective tissue disorders) | 1 (1) — Recovery after surgery took longer than the time frame the surgeon gave. Patient struggled to move fingers and wrist significantly post-surgery
Complex Regional Pain Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient experiences significant pain when lifting any heavy object and has ongoing weakness in affected hand/wrist
Pain in wrist (Musculoskeletal and connective tissue disorders) | 2 (2) — 1. Patient's wrist was still quite painful, causing some difficulty sleeping at night and has minimal range of movement - wrist was slightly swollen, slightly hypersensitive thumb with some occasional pins and needles 2. Pain and discomfort in wrist
Reduced ROM (Musculoskeletal and connective tissue disorders) | 5 (5) — 1. Slightly reduced ROM-wrist flexion and some resistance when making a tight fist 2. Reduced ROM in wrist 3. Slight reduced range of motion- hand not flat during yoga 4. Stiffness, reduced ROM and some pain 5. Reduced wrist ROM affecting activities
Pain when lifting heavy objects (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient struggles with pain when lifting heavy objects (more than 5kg) and with repeated movements like using a tin opener or using bathroom tissue. Patient avoids these activities.
Occasional pain and slightly reduced ROM (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient since operation gets occasional pain and slight reduced ROM, only at it's worse during cold weather. The pain rarely affects the patient.
Numbness (Nervous system disorders) | 1 (1) — Patient experiences numbness in thumb, index & middle fingers which is related to the nerve dysfunction
Swollen wrist (Musculoskeletal and connective tissue disorders) | 1 (1) — Swollen wrist with a globally reduced range of motion which results to the hand movement stiffness
Polymyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain post operatively leading to prolonged stay. Background of Polymyalgia which can often predispose to pain control issues. Difficult to say if pain from swelling of original fracture of from procedure.
Shooting nerve pain in wrist (Nervous system disorders) | 1 (1) — Patient experiences shooting/nerve pain in wrist when completing certain tasks like using a bathroom tissue. Does not occur often but can be really painful
Stitches opened (Skin and subcutaneous tissue disorders) | 1 (1) — Patient's stitches/wound opened up the day after surgery - bleeding inside the cast. Went t back to hospital to have her wound re-dressed and re-cast.
Bones moving forward (Injury, poisoning and procedural complications) | 1 (1) — Plate has not stopped the bones from moving forward
Tingling sensation (Skin and subcutaneous tissue disorders) | 2 (2) — 1. Patient experiences tingling sensation when touching the skin over the plate 2. Patient experiences regular nerve pain/twinges, and pins & needles
Clicking and minor weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient experiences clicking in wrist when moving and some minor weakness when lifting heavy objects
Thicker wrist (Product Issues) | 1 (1) — Patient's operated wrist is thicker than other (non-operated) wrist
Plate pincing nerve (Product Issues) | 1 (1) — Patient is complaining of the plate pinching a nerve in wrist causing issues with thumb (stiffness and poor flexibility)
Loss of power and grip strenght (Musculoskeletal and connective tissue disorders) | 4 (4) — 1. Small amount of loss of power & grip strength 2. Reduced grip strength-doesn't impact activities 3. Reported lower grip strength in affected hand/wrist 4. Reduced strength and infrequent pain-worse/intense when using wrist for certain activities
Concurring spinal injuries (Injury, poisoning and procedural complications) | 1 (1) — Patient had delayed discharge due to concurring spinal injuries
Collapse at fracture site (Product Issues) | 1 (1) — Collapse at fracture site resulting in metalwork removal (plate and screws)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back pain/nerve pain in back that sometimes affects both arms
Stiffness and irritation caused by the plate (Product Issues) | 2 (2) — 1. Patient experienced stiffness of wrist (no pain) and irritation cause by the plate 2. Patient experiences significant stiffness and reduced range of motion resulting in the plate being removed. Stiffness remains after device removal
Dull ache (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient experiences dull ache in wrist, this pain can prevents patient from doing push-ups and from writing for extended periods of time
Wrist weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Patient experiences some wrist weakness
Enlarged scar (Skin and subcutaneous tissue disorders) | 1 (1)
Pins and needles feeling (Nervous system disorders) | 2 (2) — 1. Patient experiences ongoing pins and needles in affected hand/wrist 2. Patient experiencing pins & needles in wrist, extending to forearm for the last 1-2 years
Pain combined with stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) — 1. Patient has ongoing pain/aches in wrist, stiffness and reduced grip strength making majority of activities more difficult 2. Patient gets pain when performing repeated wrist movements, has increased stiffness & reduced ROM when twisting wrist
Pain when performing repeated wrist movements (Musculoskeletal and connective tissue disorders) | 1 (1)
Reduced strength (Musculoskeletal and connective tissue disorders) | 2 (2) — 1. Patient has reduced level of strength in left hand 2. Patient's wrist fatigues quickly and loses strength during use. The patient also experiences regular ongoing pain in wrist
Inpatient fall (Injury, poisoning and procedural complications) | 1 (1) — Inpatient fall sustaining skull fracture with concurrent subdural hematoma - longer admission

LIMITATIONS AND CAVEATS:
The limitations of this study are that it was retrospective, over the pandemic and required extensive hours of discussion and contacting of patients which took extended time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT04653051/Prot_SAP_000.pdf